CLINICAL TRIAL: NCT07063394
Title: Evaluation of the Efficacy of Virtual Reality as a Therapeutic Method to Reduce Opioid Consumption in Postoperative Cardiac and Thoracic Surgery
Brief Title: Evaluation of Virtual Reality for Reducing Opioid Use After Cardiac and Thoracic Surgery
Acronym: VR-Opioid-Post
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Filomena R B G Galas (Other Government)
Responsible Party: Sponsor-Investigator, Filomena R B G Galas, Filomena Regina Gomes Barbosa Galas, Instituto do Coracao
Organization: Instituto do Coracao (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6.889.108; 6.889.108 (Other: Plataforma Brasil)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Heart Surgery; Thoracic Surgery; Opioid; Virtual Reality; Pain
Keywords: Heart surgery; Thoracic Surgery; Opioid; Virtual Reality; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, single-center, parallel-group trial with three arms. Participants undergoing elective cardiac or thoracic surgery will be randomized in a 1:1:1 ratio to receive: (1) standard postoperative care plus virtual reality (VR) with interactive games and/or passive imagery; (2) standard care plus VR with passive contemplative imagery only; or (3) standard postoperative care alone (control). The VR intervention will be administered over five consecutive postoperative days, with three supervised sessions per day, each lasting 30 to 45 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Participants in Group 1 will receive standard postoperative care plus virtual reality (VR) therapy using both interactive games and passive imagery. The goal is to reduce opioid consumption and improve recovery through immersive distraction. VR sessions will be held three times daily, lasting 30-45 minutes each, for five consecutive postoperative days or until discharge. Games such as Fruit Ninja 2, Beat Saber, and Oculus First Contact offer stimulating experiences, while passive content from YouTube VR provides relaxing visual environments. Patients will be trained to operate the VR device and choose content based on their preference. All sessions will be supervised by the study team to ensure proper use and maximize therapeutic effect.
  Interventions: Device: Group 1
- Group 2 (Experimental): Participants in Group 2 will receive standard postoperative care plus virtual reality (VR) therapy focused solely on passive imagery for distraction. VR sessions will occur three times daily, each lasting 30-45 minutes, for five consecutive postoperative days or until discharge. Patients will view calming, immersive content-such as nature scenes and relaxing landscapes-available on platforms like YouTube VR. These experiences aim to reduce opioid consumption and improve recovery by decreasing pain perception. Participants will be trained to use the device and guided by the study team, who will supervise each session to ensure proper use and maximize therapeutic effect.
  Interventions: Device: Group 2
- Group 3 (No Intervention): Participants in Group 3 will serve as the control group, receiving standard postoperative care without virtual reality (VR) intervention. Standard care includes institutional pain management protocols, such as the use of opioids and non-opioid analgesics after cardiac or thoracic surgery. No immersive or distraction-based technologies will be provided. This group serves as a baseline for comparison with the VR groups (Groups 1 and 2), enabling evaluation of the impact of VR on opioid consumption, pain perception, and recovery outcomes. Data from Group 3 will help assess the added value of VR as a complementary tool in postoperative care.

INTERVENTIONS:
Device: Group 1 — Patients in Group 1 will receive standard anesthesia protocol combined with interactive and immersive Virtual Reality (VR) therapy. This includes both engaging in interactive games that require cognitive and motor tasks, such as slicing objects or solving puzzles, and watching immersive 360-degree videos featuring calming environments like natural landscapes. The VR sessions are designed to distract patients from pain perception and reduce anxiety. The intervention will be administered for 3 sessions per day, each lasting 30-45 minutes, over 5 consecutive postoperative days.
  Arms: Group 1
Device: Group 2 — Patients in Group 2 will receive standard anesthesia protocol combined with passive Virtual Reality (VR) therapy. This involves the use of a VR headset to watch immersive 360-degree videos, such as tranquil natural landscapes or underwater scenes, designed to promote relaxation and reduce anxiety. The VR sessions do not require active participation, allowing patients to passively observe calming environments. The intervention will be administered for 3 sessions per day, lasting 30-45 minutes each, over 5 consecutive postoperative days.
  Arms: Group 2

SUMMARY:
This clinical trial aims to evaluate the efficacy of virtual reality (VR) as an adjunctive therapeutic method to reduce opioid consumption during the postoperative period of cardiac and thoracic surgeries. It is a single-center, prospective, randomized trial that will include 60 patients aged 16 to 40 undergoing surgeries such as valve replacements, pulmonary decortication, thoracic sympathectomies, and video-assisted thoracic procedures. Patients will be randomized into three groups:

Group 1: Standard anesthesia protocol combined with interactive VR therapy using games like Fruit Ninja 2, Beat Saber, and Oculus First Contact, as well as passive contemplation of immersive virtual environments (Blue Planet, Wander).

Group 2: Standard anesthesia protocol combined with VR therapy focusing solely on passive imagery, such as immersive 360° videos available on YouTube VR.

Group 3 (Control): Standard anesthesia protocol without any VR intervention.

The VR intervention will occur in three daily sessions lasting 30-45 minutes each, over the first five postoperative days or until hospital discharge, whichever comes first. Training in VR equipment usage and full supervision by the study team will be provided throughout all sessions.

Primary Objective:

The primary goal is to reduce total opioid consumption, measured through medical prescriptions and patient-controlled analgesia (PCA) pump usage. Pain control will be assessed using the Visual Analogue Scale (VAS).

Secondary Objectives:

Evaluate the incidence of postoperative nausea and vomiting (PONV).

Measure the duration of mechanical and non-invasive ventilation.

Assess the length of stay in the ICU and the total hospital stay.

Record the occurrence of paralytic ileus.

Evaluate patient satisfaction.

Assess cognitive status using the Mini-Mental State Examination (MMSE).

Rationale:

Postoperative pain following cardiac and thoracic surgeries is commonly treated with opioids, which are associated with adverse effects such as respiratory depression, nausea, vomiting, constipation, and risk of dependency. Virtual reality offers an innovative approach to pain management by creating immersive environments that serve as cognitive distractions. This immersive distraction modulates pain perception, reduces anxiety, and enhances overall well-being. Prior studies have shown that VR can effectively reduce pain perception and improve patient satisfaction, supporting its potential as a non-pharmacological adjunct in various clinical contexts.

Methods:

Participants will undergo standardized surgical and anesthetic protocols at the Instituto do Coração (InCor) of the Hospital das Clínicas at the University of São Paulo. Clinical and demographic data will be collected, including opioid consumption, VAS pain scores, ventilatory parameters, and other relevant recovery indicators. Statistical analyses will include descriptive statistics, univariate comparisons, and multivariate logistic regression to identify significant associations between the interventions and outcomes. Analyses will be performed using SPSS, with statistical significance set at p < 0.05.

Anticipated Outcomes:

The study anticipates that VR will significantly reduce postoperative opioid consumption, enhance pain control, and improve patient satisfaction. Additionally, patients exposed to VR may experience shorter hospital stays, reduced side effects, and better overall recovery metrics. If proven effective, VR could serve as a scalable, cost-effective, and safe complement to traditional postoperative pain management strategies, especially in populations where minimizing opioid use is a clinical priority.

Ethical Considerations:

DETAILED DESCRIPTION:
Title:

Evaluation of Virtual Reality as a Therapeutic Method for Reducing Opioid Consumption in Postoperative Pain Management after Cardiac and Thoracic Surgeries

Introduction and Background:

Pain management is one of the most significant challenges in postoperative care, particularly in patients undergoing major surgeries such as cardiac and thoracic procedures. Effective pain control is essential not only for the comfort and well-being of the patient but also for improving surgical outcomes, reducing complications, and minimizing recovery times. Traditionally, postoperative pain is managed with pharmacological interventions, particularly opioids. While opioids are highly effective in controlling acute pain, their use comes with several drawbacks. These include adverse effects such as respiratory depression, nausea, vomiting, and constipation, as well as the potential for opioid dependence, tolerance, and addiction. Additionally, the overuse of opioids contributes to the global opioid crisis, emphasizing the need for alternative pain management strategies.

Recent advancements in non-pharmacological interventions have highlighted virtual reality (VR) as a promising tool for pain management. VR employs immersive environments to engage the patient's sensory and cognitive faculties, thereby reducing the perception of pain. The mechanism is based on distraction, which modulates the patient's attention away from nociceptive stimuli. VR also triggers the release of endorphins and other neurotransmitters that enhance mood and reduce pain perception. These combined effects make VR an appealing adjunct to traditional pain management techniques, especially in settings where minimizing opioid use is critical.

Study Objectives:

The primary goal of this study is to evaluate the efficacy of VR as an adjunctive therapeutic method to reduce opioid consumption during the postoperative period of cardiac and thoracic surgeries. Secondary objectives include assessing its impact on various recovery metrics such as pain scores, nausea and vomiting, duration of mechanical ventilation, length of ICU and hospital stays, cognitive status, and overall patient satisfaction.

Primary Objective:

To measure the reduction in total opioid consumption in patients using VR as an adjunctive therapy during the first five postoperative days.

Secondary Objectives:

Evaluate the incidence of postoperative nausea and vomiting (PONV)

Assess the duration of mechanical ventilation and non-invasive ventilation

Determine the length of stay in the intensive care unit (ICU) and overall hospital stay

Investigate the occurrence of paralytic ileus

Measure patient satisfaction with the intervention

Evaluate cognitive status using the Mini-Mental State Examination (MMSE)

Record pain scores at rest and during movement using the Visual Analogue Scale (VAS)

Study Design:

This is a prospective, randomized, open-label, single-center clinical trial conducted at the Instituto do Coração (InCor) of the Hospital das Clínicas, São Paulo, Brazil. A total of 60 patients, aged 16 to 40, will be enrolled and randomized into three groups in a 1:1:1 ratio.

Participant Groups:

Group 1 (Interactive VR): Participants will use VR devices featuring interactive games (Fruit Ninja 2, Beat Saber, Oculus First Contact) or passive imagery (Blue Planet, Wander) for immersive distraction.

Group 2 (Passive VR): Participants will use VR devices to view passive imagery and relaxing videos, including 360° nature scenes available via YouTube VR, designed to induce a calming and visually engaging experience.

Group 3 (Control): Participants will receive standard institutional postoperative pain management protocols, without the use of any VR intervention.

Intervention Protocol:

The VR therapy will commence on the first postoperative day and will consist of three daily sessions of 30-45 minutes each, continuing for five consecutive days or until hospital discharge, whichever occurs first. Patients will be trained to use the VR equipment and will receive assistance to select appropriate content based on group allocation. All sessions will be supervised by the study team to ensure proper use and to maximize the therapeutic potential of the intervention.

In Group 1, participants will be allowed to choose between engaging in cognitively and physically interactive games or contemplative immersive environments. Group 2 participants will view relaxing visual content only, such as underwater scenes and natural landscapes. No VR devices or immersive tools will be offered to the control group.

Inclusion Criteria:

Patients aged 16 to 40 years

Undergoing elective cardiac or thoracic surgeries, including valve replacements, pulmonary decortication, thoracic sympathectomies, and video-assisted thoracic surgeries

Cognitive score of ≥25 on the Mini-Mental State Examination (MMSE)

Exclusion Criteria:

Visual impairments or severe motor limitations

Cognitive deficits (MMSE ≤ 24)

Claustrophobia or spatial disorientation

Vestibular disorders (e.g., severe motion sickness)

Infectious or contagious diseases

Outcome Measures:

Primary Outcome: Total opioid consumption over the five-day postoperative period, assessed via medical prescriptions and PCA pump usage.

Secondary Outcomes:

Pain intensity using the Visual Analogue Scale (VAS) at rest and during movement

Incidence of postoperative nausea and vomiting (PONV)

Duration of mechanical and non-invasive ventilation

ICU and hospital length of stay

Occurrence of paralytic ileus

Patient satisfaction scores

Cognitive performance assessed by MMSE

Data Collection and Analysis:

Data will be collected from electronic health records and include demographics, clinical variables, pain scores, analgesic prescriptions, ventilatory parameters, and hospitalization data. Statistical analysis will include descriptive statistics, univariate comparisons, and multivariate logistic regression models to identify significant associations between the intervention and outcomes. All analyses will be conducted using SPSS software, with significance set at p < 0.05.

Safety and Ethical Considerations:

This study has been approved by the institutional ethics committee and adheres to local and international ethical standards. Informed consent will be obtained from all participants before enrollment. Privacy and confidentiality of data will be ensured throughout the study. Potential adverse effects from VR use, such as cybersickness or visual discomfort, will be minimized through pre-session training, proper hygiene, time-limited use, and supervision during each session.

Anticipated Benefits:

The study anticipates that VR use will result in reduced opioid consumption, lower pain intensity, improved cognitive outcomes, and higher levels of patient satisfaction. VR may also reduce the incidence of side effects commonly associated with opioid use. These benefits could help validate VR as an effective, low-risk, and scalable complementary therapy for pain control in the postoperative setting.

Conclusion:

This trial seeks to assess the feasibility and efficacy of incorporating VR into standard postoperative care for patients undergoing cardiac and thoracic surgery. By promoting immersive distraction and reducing reliance on opioids, VR may enhance recovery, shorten hospital stays, and improve the overall patient experience. If successful, this model may be expanded to other surgical contexts and support broader integration of non-pharmacological tools in multimodal analgesia strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective cardiac or thoracic surgeries at the Heart Institute (InCor) of the Hospital das Clínicas of the University of São Paulo.
* Eligible thoracic surgeries include: pulmonary decortication, thoracic sympathectomy, video-assisted thoracoscopic surgery (VATS), pulmonary biopsy, and pectus excavatum repair using the Nuss procedure.
* Patients aged between 16 and 40 years.
* Preserved cognitive function, indicated by a Mini-Mental State Examination (MMSE) score of ≥ 25.

Exclusion Criteria:

* Visual impairments.
* Cognitive impairment (MMSE ≤ 24).
* Severe upper limb motor limitations.
* Claustrophobia.
* Spatial disorientation.
* Motion sickness or vestibular disorders.
* Infectious or contagious diseases.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Opioid Consumption | From the end of surgery up to 5 days after surgery
  Measured by the total amount of opioids administered postoperatively

SECONDARY OUTCOMES:
Occurrence of Nausea and Vomiting | Within 5 days after surgery
  Frequency of postoperative nausea and vomiting episodes
Length of ICU Stay | Within 5 days after surgery
  Number of days spent in the ICU
Length of Hospital Stay | Within 30 days after surgery
  Number of days hospitalized
Length of Mechanical Ventilation | Within 5 days after surgery
  Hours of mechanical ventilation
Length of Non-Invasive Ventilation | Within 5 days after surgery
  Hours of non-invasive ventilation
Occurrence of Paralytic Ileus | Within 5 days after surgery
  Presence of paralytic ileus postoperatively
Patient Satisfaction | Within 5 days after surgery
  Assessed using a standardized satisfaction scale
Postoperative Pain | Within 5 days after surgery
  Assessed using the Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kodvavi MS, Asghar MA, Ghaffar RA, Nadeem I, Bhimani S, Kumari V, Rabbani A, Iqbal M, Naeem R, Nasir AM, Hassan SS, Ghazni MS. Effectiveness of virtual reality in managing pain and anxiety in adults during periprocedural period: a systematic review and meta-analysis. Langenbecks Arch Surg. 2023 Aug 9;408(1):301. doi: 10.1007/s00423-023-03046-5. PMID 37556082
- [Background] Lind A, Ahsan M, Totzeck M, Al-Rashid F, Haddad A, Dubler S, Brenner T, Skarabis A, El Gabry M, Rassaf T, Janosi RA. Virtual reality-assisted distraction during transcatheter aortic valve implantation under local anaesthesia: A randomised study. Int J Cardiol. 2023 Sep 15;387:131130. doi: 10.1016/j.ijcard.2023.131130. Epub 2023 Jun 22. PMID 37355243